CLINICAL TRIAL: NCT00109382
Title: Fast Assessment of Stroke and Transient Ischemic Attack to Prevent Early Recurrence (FASTER)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Stroke Consortium (CSC) (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: CSP-100
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2007-06

CONDITIONS: Transient Ischemic Attack; Stroke
Keywords: Transient Ischemic Attack; Stroke; Stroke Prevention; Recurrence; Neuroprotection; Antiplatelet Therapy; Statins
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Recurrence | interventions — Aspirin; Clopidogrel; Simvastatin

INTERVENTIONS:
Drug: Aspirin
Drug: Clopidogrel
Drug: Simvastatin

SUMMARY:
Current management of patients with TIA (transient ischemic attack) or minor stroke includes the prompt investigation and treatment in the days and weeks after the event. However, new evidence shows patients are at the highest risk of stroke in the first few days after the TIA, with 50% of strokes which happen in the three months following TIA occurring within 48-72 hours. To date, there is no evidence to guide physicians on how to safely reduce this risk.

The FASTER trial is focusing on the initial period of high risk, starting patients on stroke prevention treatments in the hours following a TIA or minor stroke. The drugs to be tested have been shown to be effective in the similar setting of cardiology, reducing recurrent cardiac events in patients with unstable angina when commenced with the same speed after an event.

All patients will be on aspirin. The trial will see if adding another drug, clopidogrel, has an additional benefit in reducing the number of strokes after TIA or minor stroke within three months of TIA or minor stroke. It will also look if the very early introduction of simvastatin, a cholesterol lowering therapy, reduces stroke after TIA or minor stroke, both by itself and in addition to clopidogrel. The final aim of the trial is to ensure that these treatments are safe to be used in this population of patients.

DETAILED DESCRIPTION:
The Fast Assessment of Stroke and Transient ischemic attack to prevent Early Recurrence (FASTER) is a randomized clinical trial designed to investigate the effect of hyper-acute initiation of stroke prevention treatments in patients with a minor stroke or transient ischemic attack (TIA).

This group of individuals has been recognized as being at high risk of recurrent events. Johnston et al. (2000) were the first to suggest that the risk of stroke after TIA was front-loaded in the first few days. This has been confirmed elsewhere with Lovett et al. (2003) having shown in the Oxfordshire Community Stroke Project that the 7-day risk of recurrent stroke was 8.6%, and a 30-day risk of 12.0%. These findings are similarly found in the Oxford Vascular Study; 8.0% and 11.5% respectively for a recurrent event (Coull et al., 2004). The NASCET (North American Symptomatic Carotid Endarterectomy Trial) study also supports the finding of high risk of early recurrent stroke. 8.5% of patients with a hemispheric TIA suffered a recurrent stroke within one week rising to 20% at 90-days (Eliasziw et al., 2004). This data suggest that patients with carotid stenosis are at the highest risk of early recurrent stoke.

Only one in four patients with acute ischemic stroke presenting within three hours of symptom onset are being treated with t-PA (Barber et al., 2001). The most common reason for exclusion from treatment is that a patient's deficit will be too mild for treatment or will have completely resolved thereby not meriting the risks of treatment with tPA. These are the patients that have a higher risk of early recurrence. The clinical imperative is to identify hyper-acute treatment strategies to minimize that risk.

FASTER is a double blind, randomized controlled trial with a 2x2 factorial design with patients followed for 90-days. Patients will be randomized within 24 hours of symptom onset to one of four possible treatment arms:

* Aspirin
* Aspirin and Clopidogrel
* Aspirin and Simvastatin
* Aspirin and Clopidogrel and Simvastatin

Study Hypotheses

A. A rapid commencement of clopidogrel plus aspirin within 24 hours of acute TIA or minor stroke is more effective than aspirin in reducing the 90-day risk of stroke by an absolute difference of 2%.

B. A rapid commencement of simvastatin plus aspirin within 24 hours of acute TIA or minor stroke is more effective than aspirin in reducing the 90-day risk of stroke by an absolute difference of 2%.

C. A rapid commencement of clopidogrel plus aspirin plus simvastatin within 24 hours of acute TIA or minor stroke is more effective than aspirin alone in reducing the 90-day risk of stroke by an absolute difference of 4%.

D. The incidence of adverse events is not different among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TIA or minor acute ischemic stroke (NIHSS < 4 at the time of randomization) who must NOT be candidates for acute thrombolysis or other acute intervention indicated as the current standard of care
* Aged 40 years or older
* Patients with: (a) weakness at time of TIA/minor stroke and/or language disturbance at time of TIA/minor stroke and; (b) duration of neurological deficit (TIA) > 5 minutes
* Patients can be randomized within 24 hours of symptom onset. Symptom onset is defined by the "last seen well" principle
* Patients must have provided written, informed consent to participate in the FASTER trial.

Exclusion Criteria:

* Patients with pure sensory symptoms, pure vertigo or dizziness, pure ataxia or pure visual loss
* Patients for whom thrombolysis or other acute intervention is indicated as the current standard of care
* Patients who are currently on statin therapy, antiplatelet therapy (not including aspirin), or long-term non-steroidal anti-inflammatory drugs (NSAIDs but not COX inhibitors), or anticoagulation
* Patients who in the opinion of the site Investigator, should be commenced on statin therapy
* Patients with neurological deficit due to intracranial hemorrhage (intracranial hemorrhage, subarachnoid hemorrhage, subdural hematoma, epidural hematoma), tumor, infection or any finding not consistent with acute brain ischemia as the cause of presenting symptoms
* Presumed cardiac source of embolus (e.g. atrial fibrillation, prosthetic cardiac valve, known/suspected endocarditis)
* Patient with a concomitant acute coronary syndrome (acute myocardial infarction or unstable angina)
* Modified Rankin Score 3 or more (pre-morbid historical assessment)
* Patients in whom the qualifying event was due to a complication of cerebral angiography, a revascularization procedure or trauma
* Uncontrolled hypertension at baseline (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg), or malignant hypertension defined by brain plus acute organ involvement due to acute hypertension
* Women who are breast-feeding or pregnant. Women of childbearing potential must have a negative pregnancy test prior to randomization. Women of childbearing potential may still participate in the trial but must plan on not becoming pregnant during the course of the study and must practice a suitable method of birth control. If a patient becomes pregnant or begins breast-feeding during the study, both study drugs will be discontinued immediately, and the patient followed for the duration of the study
* Evidence of contraindication for use of Trial Medication: (i) serious systemic bleeding precluding antiplatelet therapy; (ii) hypersensitivity to aspirin, thienopyridine drugs (clopidogrel or ticlopidine) or statins; (iii) current or past history of renal insufficiency [serum Creatinine >150 umol]; (iv) hepatic dysfunction indicated by any or all of the following [ALT >3xULN, AST >3xULN, ALP >3xULN]; (v) thrombocytopenia [platelet count < 150 x10^9/L]; (vi) neutropenia [neutrophil count < 0.5 x10^9/L]; (vii) bleeding diathesis or coagulopathy indicated by any or all of the following [INR >1.2, PT >1.2xULN, PTT >1.2xULN]
* Life expectancy of less than 90 days
* Participation in another clinical therapeutic trial (drug or device) either concurrently or within the previous 30 days, or prior participation in FASTER
* Geographical or other factors that render follow-up impractical or that render evaluation of outcome events impossible (e.g. severe dementia). Patients may be randomized who could and are willing to complete their follow-up at a participating centre

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2003-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Any stroke at 90 days
Stroke severity

SECONDARY OUTCOMES:
Composite of stroke
Myocardial infarction
Vascular death at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alastair M Buchan, Principal Investigator — Dept of Clinical Neurosciences, University of Calgary; James Kennedy, Study Director — Nuffield Dept of Clinical Medicine, University of Oxford
Locations (18):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Canada (17):
  - Foothills Medical Centre, Calgary, Alberta
  - Universtiy of Alberta Walter MacKenzie Health Sciences Centre, Edmonton, Alberta
  - University of Lethbridge Hospital, Lethbridge, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Centre for Stroke Research, Victoria, British Columbia
  - St. John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth ll Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Women's Health Centrre, Toronto, Ontario
  - St. Mike's Hospital, Toronto, Ontario
  - Toronto Western Hospital -University Health Network, Toronto, Ontario
  - Chicoutimi Hospital, Chicoutimi, Quebec
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

REFERENCES:
- [Background] Palumbo V, Eliasziw M, Buchan AM, on behalf of the FASTER Investigators. Urgent Stroke Imaging is also Feasible for Secondary Prevention Trial. 28th International Conference on Stroke and Cerebral Circulation, American Heart Association Stroke Conference. Clinical Trials Abstract. Accepted as Poster Presentation. 2003
- [Background] Kennedy J, Eliasziw M, Buchan AM on behalf of the FASTER Collaborators. The Fast Assessment of Stroke and Transient ischemic attack to prevent Early Recurrence (FASTER) Trial. 28th International Conference on Stroke and Cerebral Circulation, American Heart Association Stroke Conference. Clinical Trials Abstract. http://www.strokeconference.org/sc_includes/pdfs/CTP24.pdf Accepted as Poster Presentation. 2003
- [Background] Kennedy J, Eliasziw M, Hill MD, Buchan AM. The Fast Assessment of Stroke and Transient ischemic attack to prevent Early Recurrence (FASTER) Trial. Seminars in Cerebrovascular Diseases and Stroke, March 2003 Ed. J. Biller. Vol 3/1 pp 25-30. 2003
- [Background] Kennedy J, Eliasziw M, Buchan AM on behalf of the FASTER Investigators. The Fast Assessment of Stroke and Transient ischemic attack to prevent Early Recurrence (FASTER) Trial. 29th International Conference on Stroke and Cerebral Circulation, American Heart Association Stroke Conference. Clinical Trials Abstract. Accepted as Poster Presentation. 2004
- [Background] Kennedy J, Ma C, Buchan AM. FASTER prevention, fastest neuroprotection. Pharmacology of Cerebral Ischemia, Proceedings of the Marburg Conference 2004. Ed. J Krigelstein. (In Press)
- [Background] Kennedy J, Buchan AM on behalf of the FASTER Investigators. The Fast Assessment of Stroke and Transient ischemic attack to prevent Early Recurrence (FASTER) Trial. 30th International Conference on Stroke and Cerebral Circulation, American Heart Association Stroke Conference. Clinical Trials Abstract. Accepted as Poster Presentation. 2005
- [Background] Eliasziw M, Kennedy J, Hill MD, Buchan AM, Barnett HJ; North American Symptomatic Carotid Endarterectomy Trial Group. Early risk of stroke after a transient ischemic attack in patients with internal carotid artery disease. CMAJ. 2004 Mar 30;170(7):1105-9. doi: 10.1503/cmaj.1030460. PMID 15051694
- [Derived] Kennedy J, Hill MD, Ryckborst KJ, Eliasziw M, Demchuk AM, Buchan AM; FASTER Investigators. Fast assessment of stroke and transient ischaemic attack to prevent early recurrence (FASTER): a randomised controlled pilot trial. Lancet Neurol. 2007 Nov;6(11):961-9. doi: 10.1016/S1474-4422(07)70250-8. Epub 2007 Oct 10. PMID 17931979